CLINICAL TRIAL: NCT04471181
Title: Greek Ruptured Aneurysm Endovascular Repair Study
Brief Title: Greek Study for Endovascular Repair of Ruptured Abdominal Aortic Aneuryms
Acronym: GRAND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kostantinos Papazoglou (Other)
Collaborators: Medtronic (Industry); Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor-Investigator, Kostantinos Papazoglou, Professor in Vascular surgery, Ippokrateio General Hospital of Thessaloniki
Organization: Ippokrateio General Hospital of Thessaloniki (Other)
Other Study IDs: GRAND study
Record Dates: First submitted 2020-07-05; First posted 2020-07-15 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Rupture, Aortic; Aneurysm, Abdominal Aortic; Aneurysm, Ruptured
Keywords: Ruptured Abdominal Aortic Aneurysm; Endovascular Repair
MeSH Terms: conditions — Aortic Rupture; Aortic Aneurysm, Abdominal; Aneurysm, Ruptured

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- All patients with ruptured abdominal aortic aneurysms: All patients will undergo CTA to confirm the diagnosis. The use of balloon for aortic clamp in case of haemodynamic instability can be used.
  All patients included in the research study must undergo standard EVAR with a bifurcated graft or an aorto-uni-iliac and a femoral to femoral crossover. In aneurysms with short proximal neck down to 4mm, or in cases where completion angiography indicates type Ia endoleak, the Heli-FX EndoAnchor system is recommended to be used, as indicated. All patients will have plain abdominal x-rays on discharge. Participants will undergo CTA in 3months and annually post-op.. In case of an adverse event before the 3 months follow up CTA, a more urgent imaging might be requested and proceed to appropriate action according to the findings.
  Interventions: Device: Endovascular repair of ruptured abdominal aortic aneurysm (EVAR) with Medtronic Endurant

INTERVENTIONS:
Device: Endovascular repair of ruptured abdominal aortic aneurysm (EVAR) with Medtronic Endurant — Endovascular repair (EVAR) of ruptured abdominal aortic aneurysms with Medtronic Endurant II, and IIs device

SUMMARY:
This will be a non-randomized, prospective, observational multi-center research study. Its purpose will be to assess the mortality and outcome of EVAR in patients with rAAA. As mentioned in the introduction, EVAR approach for ruptured bdominal aortic aneurysms is nowdays common clinical practice in many vascular centers , and the main treatment option in Hippokrateio General hospital. The same applies in all future participating vascular centers.

DETAILED DESCRIPTION:
Ruptured abdominal aortic aneurysms (rAAAs) remain one of the most emergent medical events, with over 90% mortality if left untreated and a prevalence of a minimum 45 patients per 1000000 population. The 30 day mortality for emergency open repair has remained at around 50%, and there is no consistent improvement in the outcome of the open technique over time. Since its development, endovascular aneurysm repair (EVAR), has been increasingly used even in the emergency setting.

So far there have been 4 randomized controlled trials, comparing EVAR versus open repair for rAAA. The first was a small trial from Nottingham followed by the Dutch trial AJAX and the French ECAR. The last and biggest trial with 613 patients was the UK IMPROVE trial. All these trials showed non inferiority of EVAR, but failed to prove benefit for EVAR with respect to 30 day mortality. Furthermore two meta-analysisof the above RCTs, stated again, that 30 and 90 day mortality is similar between EVAR and open surgery, with the exception of women having a better outcome with an endovascular approach.

On the contrary, multiple observational studies and registries showed even a 50% risk reduction in mortality with EVAR. There has been huge critique and discussion of the results in IMPROVE trial, in which 10% of patients crossed over to the non-allocated treatment group. In both groups, patients who were treated with EVAR had a mortality of 25%, significantly lower than those who received open surgery (38%). Furthermore, two recent published studies that compared mortality of rAAA between Sweden, USA and UK, came to the conclusion that mortality is lower in centers that accept a large number of cases with rAAA, mostly treated with EVAR. There is an argument that these encouraging results are subject of bias, since there is patient selection according to haemodynamic stability and aortic morphology. A valid counter argument stated by Lachat and colleagues is that EVAR for rAAA in their center, in the moderate risk, stable patient with favourable anatomy (aortic neck length >10mm) has a reduced 30 day mortality of 10%, a result never demonstrated with open repair. As EVAR evolves, new technical features of the devices may address the current limitations of the technique. In addition, the anatomic suitability obstacle for EVAR has been revoked by the PROTAGORAS study, which led to CE mark for a commercial stent graft system, allowing treatment of aortic neck lengths as small as 2mm with the use of chimney technique. The authors in the IMPROVE trial acknowledge the fact that: "The suitability of ruptured aneurym for EVAR is subjective and will be defined by the aortic morphology, the experience of the operator and the range of resuscitation, endovascular and anaesthetic techniques available".

It is safe to guess that haemodynamically compromised patients would benefit from a less invasive procedure, with minimum surgical exposure, if any, and local anaesthesia. There is no doubt however that for a center to adopt an EVAR only policy, poses many logistical challenges.

The aim for this research study is that an "EVAR first" approach is feasible in rAAA, even in more complex anatomies and in patients with less physiologic reserve and at the same time prove that short and midterm mortality and morbidity with EVAR is significantly lower than open repair when compared to the mortality and morbidity rates of patients receiving open repair in the latest RCT "IMPROVE". This can be achieved, with implementing a treatment alogorithm for the pre intra and post operative time, based on already established protocols and relevant international standards, with single aim to avoid the factors in patient management that contribute to mortality and morbidity. Furthermore this research study will show increased applicability of EVAR in ruptured AAAs with shorter and larger in diameter proximal neck and with angulation >60 degrees, with the implementation of EndoAnchors (HeliFX). Another aim for this research study is to identify the role of the clotting mechanism in the overall mortality and thus to distinguish patient clotting profiles that can predict or alter the outcome.

ELIGIBILITY:
Inclusion Criteria:

* All alive patients admitted with rAAA and have anatomic suitability for EVAR according to manufacturer's IFU. More accurately the anatomic criteria for the research study are :

  * Neck diameter >17mm, < 32mm
  * Angle between the suprarenal aorta and the juxtarenal aorta <60 degrees
  * Angle between the juxtarenal aorta and the long axis of the aneurysm sac <90 degrees
  * Neck length >10mm
  * Neck length <10mm down to 4mm with Heli-FX EndoAnchor system
  * Adequate aortic bifurcation diameter in case of a bifurcated graft
  * Bilateral Iliac luminal diameter >7mm

The vascular surgeon in charge will make the ultimate decision on suitability. All consecutive rAAAs treated with Endurant will be collected to avoid selection bias. No other criteria (e.g, mental illness, dementia, old age, comorbidities) will be applied to decline treatment and inclusion to the protocol. The final inclusion criterion will be that any vascular surgeon participating in the research study, must have carried out a minimum of 20 EVAR procedures for asymptomatic/symptomatic AAA. Apart from the initial 6 centers more centers can be implemented in the research study in the future.

AAA rupture will be confirmed and defined with computed tomography angiography (CTA). Rupture will be rated as free intraperitoneal rupture (free rupture), definite contrast extravasation and haematoma around the aorta (retroperitoneal rupture) and haematoma surrounding the aorta without definite contrast leak (contained rupture)

Exclusion Criteria:

* Symptomatic non ruptured AAAs will not be included even when treated as emergencies. Thoracoabdominal aneurysms and aortic dissections will also be excluded from the research study. Juxtarenal ruptured AAA treated with standard EVAR without chimney technique, outside IFU will also be excluded from the research study.However all consecutive rAAAs in the participating centers will be collected in a screening CRF to understand if this relates to rEVAR applicability.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive alive patients with true ruptured abdominal aortic aneurysm and anatomic suitability for EVAR
Sampling Method: Probability Sample
Enrollment: 157 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Mortality Rate | 30 days
  Any cause mortality after EVAR

SECONDARY OUTCOMES:
Time from rupture to diagnosis | pre-intervention
  In minutes
Time from diagnosis to intervention | pre-intervention
  In minutes
Rate of procedures converted to open repair | 24 hours post-operatively
  Any reason for conversion to open repair
Total mortality rate | 12 months post-operatively
  All cause mortality
Rate of Major Adverse Events (MAE) | 30 days, 3 months and 12 months
  MAE include :bowel ischaemia, myocardial infraction, paraplegia, renal failure, stroke, abdominal compartment syndrome, lower limb ischeamia
Rate of Endoleaks | immediately after the procedure, 3 months after the procedure, 12 months after the procedure
  Any endoleak observed
Rate of Graft related complications | 12 months after the procedure
  Any graft related complication
Fibrinogel levels | Pre-intervention, 24 hours after the procedure, 3 months after the procedure,12 months after the procedure
  Fibrinogen levels mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Kostantinos Papazoglou, Professor, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Ippokrateio General Hospital, Thessaloniki, Macedonia, Greece

IPD SHARING:
Plan to Share IPD: Yes
All IPD data that underlie results in a publication will be released by the end of the study
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: By the end of the study, until publication
Access Criteria: GDPR compatible

REFERENCES:
- [Background] IMPROVE Trial Investigators; Powell JT, Sweeting MJ, Thompson MM, Ashleigh R, Bell R, Gomes M, Greenhalgh RM, Grieve R, Heatley F, Hinchliffe RJ, Thompson SG, Ulug P. Endovascular or open repair strategy for ruptured abdominal aortic aneurysm: 30 day outcomes from IMPROVE randomised trial. BMJ. 2014 Jan 13;348:f7661. doi: 10.1136/bmj.f7661. PMID 24418950
- [Background] Hinchliffe RJ, Bruijstens L, MacSweeney ST, Braithwaite BD. A randomised trial of endovascular and open surgery for ruptured abdominal aortic aneurysm - results of a pilot study and lessons learned for future studies. Eur J Vasc Endovasc Surg. 2006 Nov;32(5):506-13; discussion 514-5. doi: 10.1016/j.ejvs.2006.05.016. Epub 2006 Aug 1. PMID 16887369
- [Background] Reimerink JJ, Hoornweg LL, Vahl AC, Wisselink W, van den Broek TA, Legemate DA, Reekers JA, Balm R; Amsterdam Acute Aneurysm Trial Collaborators. Endovascular repair versus open repair of ruptured abdominal aortic aneurysms: a multicenter randomized controlled trial. Ann Surg. 2013 Aug;258(2):248-56. doi: 10.1097/SLA.0b013e31828d4b76. PMID 23549424
- [Background] Desgranges P, Kobeiter H, Katsahian S, Bouffi M, Gouny P, Favre JP, Alsac JM, Sobocinski J, Julia P, Alimi Y, Steinmetz E, Haulon S, Alric P, Canaud L, Castier Y, Jean-Baptiste E, Hassen-Khodja R, Lermusiaux P, Feugier P, Destrieux-Garnier L, Charles-Nelson A, Marzelle J, Majewski M, Bourmaud A, Becquemin JP; ECAR Investigators. Editor's Choice - ECAR (Endovasculaire ou Chirurgie dans les Anevrysmes aorto-iliaques Rompus): A French Randomized Controlled Trial of Endovascular Versus Open Surgical Repair of Ruptured Aorto-iliac Aneurysms. Eur J Vasc Endovasc Surg. 2015 Sep;50(3):303-10. doi: 10.1016/j.ejvs.2015.03.028. Epub 2015 May 20. PMID 26001320
- [Background] van Beek SC, Conijn AP, Koelemay MJ, Balm R. Editor's Choice - Endovascular aneurysm repair versus open repair for patients with a ruptured abdominal aortic aneurysm: a systematic review and meta-analysis of short-term survival. Eur J Vasc Endovasc Surg. 2014 Jun;47(6):593-602. doi: 10.1016/j.ejvs.2014.03.003. Epub 2014 Apr 18. PMID 24746873
- [Background] Sweeting MJ, Balm R, Desgranges P, Ulug P, Powell JT; Ruptured Aneurysm Trialists. Individual-patient meta-analysis of three randomized trials comparing endovascular versus open repair for ruptured abdominal aortic aneurysm. Br J Surg. 2015 Sep;102(10):1229-39. doi: 10.1002/bjs.9852. Epub 2015 Jun 24. PMID 26104471
- [Background] Karthikesalingam A, Holt PJ, Vidal-Diez A, Ozdemir BA, Poloniecki JD, Hinchliffe RJ, Thompson MM. Mortality from ruptured abdominal aortic aneurysms: clinical lessons from a comparison of outcomes in England and the USA. Lancet. 2014 Mar 15;383(9921):963-9. doi: 10.1016/S0140-6736(14)60109-4. PMID 24629298
- [Background] Karthikesalingam A, Wanhainen A, Holt PJ, Vidal-Diez A, Brownrigg JR, Shpitser I, Bjorck M, Thompson MM, Mani K. Comparison of long-term mortality after ruptured abdominal aortic aneurysm in England and Sweden. Br J Surg. 2016 Feb;103(3):199-206. doi: 10.1002/bjs.10049. Epub 2015 Dec 1. PMID 26620854
- [Background] Vogel TR, Dombrovskiy VY, Haser PB, Graham AM. Has the implementation of EVAR for ruptured AAA improved outcomes? Vasc Endovascular Surg. 2009 Jun-Jul;43(3):252-7. doi: 10.1177/1538574408329271. Epub 2009 Jan 8. PMID 19131375
- [Background] Veith FJ, Lachat M, Mayer D, Malina M, Holst J, Mehta M, Verhoeven EL, Larzon T, Gennai S, Coppi G, Lipsitz EC, Gargiulo NJ, van der Vliet JA, Blankensteijn J, Buth J, Lee WA, Biasi G, Deleo G, Kasirajan K, Moore R, Soong CV, Cayne NS, Farber MA, Raithel D, Greenberg RK, van Sambeek MR, Brunkwall JS, Rockman CB, Hinchliffe RJ; RAAA Investigators. Collected world and single center experience with endovascular treatment of ruptured abdominal aortic aneurysms. Ann Surg. 2009 Nov;250(5):818-24. doi: 10.1097/SLA.0b013e3181bdd7f5. PMID 19809296
- [Background] Papazoglou K, Mallios A, Rafati F, Zambas N, Karkos C. Endovascular treatment of ruptured abdominal aortic aneurysms with the Endurant device. Ann Vasc Surg. 2013 Feb;27(2):162-7. doi: 10.1016/j.avsg.2012.04.013. Epub 2012 Sep 12. PMID 22981014
- [Background] Donas KP, Torsello GB, Piccoli G, Pitoulias GA, Torsello GF, Bisdas T, Austermann M, Gasparini D. The PROTAGORAS study to evaluate the performance of the Endurant stent graft for patients with pararenal pathologic processes treated by the chimney/snorkel endovascular technique. J Vasc Surg. 2016 Jan;63(1):1-7. doi: 10.1016/j.jvs.2015.07.080. Epub 2015 Oct 23. PMID 26476671
- [Background] Mayer D, Aeschbacher S, Pfammatter T, Veith FJ, Norgren L, Magnuson A, Rancic Z, Lachat M, Horer T, Skoog P, Larzon T. Complete replacement of open repair for ruptured abdominal aortic aneurysms by endovascular aneurysm repair: a two-center 14-year experience. Ann Surg. 2012 Nov;256(5):688-95; discussion 695-6. doi: 10.1097/SLA.0b013e318271cebd. PMID 23095611
- [Background] Chaikof EL, Blankensteijn JD, Harris PL, White GH, Zarins CK, Bernhard VM, Matsumura JS, May J, Veith FJ, Fillinger MF, Rutherford RB, Kent KC; Ad Hoc Committee for Standardized Reporting Practices in Vascular Surgery of The Society for Vascular Surgery/American Association for Vascular Surgery. Reporting standards for endovascular aortic aneurysm repair. J Vasc Surg. 2002 May;35(5):1048-60. doi: 10.1067/mva.2002.123763. No abstract available. PMID 12021727
- [Background] Vu KN, Kaitoukov Y, Morin-Roy F, Kauffmann C, Giroux MF, Therasse E, Soulez G, Tang A. Rupture signs on computed tomography, treatment, and outcome of abdominal aortic aneurysms. Insights Imaging. 2014 Jun;5(3):281-93. doi: 10.1007/s13244-014-0327-3. Epub 2014 May 1. PMID 24789068
- [Background] Mell MW, Starnes BW, Kraiss LW, Schneider PA, Pevec WC. Western Vascular Society guidelines for transfer of patients with ruptured abdominal aortic aneurysm. J Vasc Surg. 2017 Mar;65(3):603-608. doi: 10.1016/j.jvs.2016.10.097. PMID 28236914
- [Result] Anjum A, von Allmen R, Greenhalgh R, Powell JT. Explaining the decrease in mortality from abdominal aortic aneurysm rupture. Br J Surg. 2012 May;99(5):637-45. doi: 10.1002/bjs.8698. PMID 22473277